CLINICAL TRIAL: NCT04806425
Title: The Cardioprotective Effect of Intralipid in Decreasing the Ischemic Insults During Off-pump Coronary Artery Revascularization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R 126/2020
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL group (Active Comparator): receive 1.5 ml /kg intralipid 20% through Central venous line after sternotomy over 1 hour
  Interventions: Drug: Intralipid
- NS group (Placebo Comparator): recieve 1.5 ml /kg normal saline 0.9% through central venous line after sternotomy over 1 hour
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intralipid — intralipid is given as a preconditioning drug during off bump coronary artery bypass grafting surgery to measure efficacy in decreasing post operative ischemia
  Arms: IL group
Drug: Placebo — normal saline is given in same volume to normal saline group over the same duration
  Arms: NS group

SUMMARY:
the aim of the study is to assess the effect of intralipid as regard efficiency in decreasing myocardial ischemia , given during preconditioning in off pump coronary artery revascularization

ELIGIBILITY:
Inclusion Criteria:

* patients between 40 to 75 undergoing off bump CABG surgery

Exclusion Criteria:

* emergency surgery
* Ejection fraction less than 50%
* redo procedures
* history of allergy to peanuts

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
ICU stay | long icu stay is considered if more than 7 days
  measuring the duration of stay in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, (Select), Egypt